CLINICAL TRIAL: NCT04787445
Title: Effects of Pulmonary Hypertension Therapy in Atypical Pulmonary Arterial Hypertension: An Exercise Hemodynamic Study (TAPH Study)
Brief Title: Effects of Pulmonary Hypertension Therapy in Atypical Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Other Study IDs: 20-009542
Record Dates: First submitted 2021-02-15; First posted 2021-03-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Right Heart Catheterization
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with and without DNA will both be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to characterize the clinical and hemodynamic response of Pulmonary Arterial Hypertension (PAH) therapy in patients with atypical PAH and risk factors for left heart disease.

DETAILED DESCRIPTION:
This is an observational prospective study to better understand the clinical impact of Pulmonary Arterial Hypertension (PAH) specific therapy in patients with atypical PAH among those with risk factors for left heart disease

The study involves detailed baseline clinical evaluation prior to initiation of PAH therapy, followed by repeat clinical assessment after 6 months of medical therapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pulmonary hypertension with mean PA pressure >20 mmHg and a planned initiation of pulmonary arterial hypertension therapy
* No active treatment for precapillary pulmonary hypertension
* Ambulatory (not wheelchair/scooter dependent)
* Presence of any risk factor for left heart disease will qualify for inclusion (either atrial fibrillation, body mass index>30 kg/m2, arterial hypertension, diabetes, coronary artery disease or age>60 years)

Exclusion Criteria:

* Significant chronic obstructive pulmonary disease that is a primary contributor to symptoms in the opinion of the investigator
* Ischemia thought to contribute to dyspnea in the opinion of the investigator
* Obstructive hypertrophic cardiomyopathy
* Known infiltrative cardiomyopathy (amyloid)
* Constrictive pericarditis or tamponade
* Active myocarditis
* Complex congenital heart disease
* More than mild aortic or mitral stenosis
* Intrinsic (prolapse, rheumatic) valve disease with more than moderate mitral, tricuspid or aortic regurgitation
* Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment
* Terminal illness (other than HF) with expected survival of less than 1 year
* Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months.
* Inability to comply with planned study procedures
* Pregnancy or breastfeeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified from screening of the pulmonary hypertension clinic who are then planned for outpatient catheterization for diagnosis and management of their atypical PAH.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Describe prevalence of occult left heart disease during exercise in atypical pulmonary hypertension, as defined by pulmonary arterial wedge pressure during exercise cardiac catheterization. | Baseline Catheterization
  Pulmonary arterial wedge pressure >25 mmHg during exercise cardiac catheterization will indicate occult left heart disease.
Evaluate the therapeutic response of chronic pulmonary vasodilator therapy | 6 Month Catheterization
  Favorable pulmonary vasodilatory effect will be associated a change of > 10% reduction in pulmonary artery-pressure flow slope from baseline to 6 month catheterization

OTHER OUTCOMES:
Identify predictors on baseline exercise catheterization of subsequent exercise capacity improvement following chronic pulmonary vasodilatory therapy. | 6 Month Catheterization
  From paired exercise capacity measurements of peak VO2 from baseline to 6 month testing, patients with clinically meaningful change defined by improvement following treatment of >1 ml/kg/min will be identified. Measurements on baseline exercise catheterization, echocardiography, left atrial strain and clinical characteristics will be assessed for their ability to predict exercise capacity improvement by logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh N Reddy, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials